CLINICAL TRIAL: NCT00005645
Title: Phase II Trial of ILX295501 Administered Orally Once Weekly x 3 Repeated Every 6 Weeks in Patients With Stage III/IV Ovarian Cancer
Brief Title: ILX-295501 in Treating Patients With Stage III or Stage IV Ovarian Cancer That Has Not Responded to Previous Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Purpose: Treatment
Other Study IDs: CDR0000067825; ILEX-295501-211; CND-99-039; UCLA-9908032
Record Dates: First submitted 2000-05-02; First posted 2004-05-26 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2001-02

CONDITIONS: Fallopian Tube Cancer; Metastatic Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; liver metastases; malignant pericardial effusion; malignant pleural effusion; malignant ascites; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Neoplasm Metastasis; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Pleural Effusion, Malignant | interventions — N-(5-(2,3-dihydrobenzofuryl)sulfonyl)-N'-(3,4-dichlorophenyl)urea

INTERVENTIONS:
Drug: ILX-295501

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ILX-295501 in treating patients who have stage III or stage IV ovarian cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response in patients with refractory stage III or IV ovarian epithelial cancer treated with ILX-295501. II. Determine the number of patients with at least 50% decrease in CA125 when treated with this regimen. III. Determine the time to tumor progression, overall survival, and toxicity profile in this patient population treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive oral ILX-295501 once weekly for 3 weeks. Treatment repeats every 6 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed at 1 month and then every 3 months until death.

PROJECTED ACCRUAL: A total of 30-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III or IV ovarian epithelial cancer, including fallopian tube and extraovarian carcinoma Cytological confirmation in the presence of clear clinical and radiological features of disease allowed Refractory to at least two prior chemotherapy regimens for advanced or metastatic disease At least one taxane/platinum containing regimen with or without one topotecan regimen Recurrent or progressive disease while on or within 6 months of last therapy regimen Must have progressed on or within 3 months of receiving topotecan as last therapy regimen Measurable disease outside previously irradiated field OR Objective evidence of disease progression if within previously irradiated field CA 125 at least 35 units/mL No CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST and ALT no greater than 3 times ULN (no greater than 5 times ULN if liver metastases present) Albumin greater than 2.5 g/dL Renal: Creatinine no greater than ULN Other: No known hypersensitivity to sulfa compounds No known glucose-6-phosphate dehydrogenase deficiency No active or uncontrolled infection No other malignancy within the past 2 years No other severe disease including neurologic or psychiatric disorders that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy and recovered No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy, excluding contraceptives or corticosteroids Radiotherapy: See Disease Characteristics Prior radiotherapy to less than 25% bone marrow allowed No prior whole pelvic radiotherapy At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: At least 4 weeks since prior major surgery and recovered Other: At least 4 weeks since prior investigational agents No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-05

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Cook, RN, Study Chair — Genzyme, a Sanofi Company
Locations (8):
- United States (8):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Mercy Medical Center, Inc., Baltimore, Maryland
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Billings Oncology Associates, Billings, Montana
  - St. Vincents Comprehensive Cancer Center, New York, New York
  - Sarah Cannon-Minnie Pearl Cancer Center, Nashville, Tennessee
  - Virginia Mason Medical Center, Seattle, Washington